CLINICAL TRIAL: NCT00824213
Title: Pilot Project: Fast Whole-body Spect Scanning to Improve the Detection of Bone Metastases in Patients With Diagnosed Cancer
Status: Completed | Type: Observational
Sponsor: University of British Columbia (Other)
Responsible Party: Dr. Anna Celler, University of British Columbia
Other Study IDs: H08-01640
Record Dates: First submitted 2009-01-14; First posted 2009-01-16 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-03

CONDITIONS: Bone Metastases
Keywords: Whole Body SPECT imaging

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The investigators propose to investigate the performance of the image reconstruction software with resolution recovery correction for bone SPECT studies. The investigators estimate that in only 30 minutes, using this new technique of collimator de-blurring, one could perform a fully 3-dimensional SPECT whole-body bone study, essentially obviating the necessity for doing planar bone studies.

In the scope of the proposed project, the investigators group aims to test the hypothesis that one can perform a Tc-99m whole-body SPECT study in the same time as a regular routine planar bone study, with greater localization accuracy, and greater lesion detection.

To establish a "gold standard" necessary to assess the performance of the SPECT bone scans, the investigators will compare number of malignant lesions detected in patients who are proven to have metastatic skeletal bone lesions on PET F-18 whole-body scans, with whole-body Tc-99m SPECT lesions. The investigators also propose to compare the detection of SPECT scans with standard planar bone scans. This will allow for two major comparisons (a) the accuracy of SPECT bone studies compared to planar bone studies, and (b) the accuracy of SPECT bone scans compared to F-18 PET studies. Most prior studies purporting to show the superiority of F-18 bone scans to Tc-99 bone scans were done only against either planar scans or a combination of planar scans and partial SPECT studies over the spine. We anticipate that F-18 bone scans, due to the higher counting statistics of PET agents, will show more lesions than SPECT, but the exact increase in sensitivity has never been compared to whole-body SPECT scans.

DETAILED DESCRIPTION:
Introduction

Bone scintigraphy (e.g. "bone scan") with Tc-99m diphosphonates is one of the most common imaging radioisotope procedures in departments of nuclear medicine worldwide, with several thousand performed every year in a busy nuclear medicine service. Despite giving fast and accurate skeletal surveys in conditions ranging from metastatic cancer, to fractures, to infection, the technology has seen little change since the early 1970's. The Anger camera remains the instrument of choice for taking serial images of a patient's skeleton, and since the late 1970's SPECT (Single Photon Emission Computed Tomography) - essentially "nuclear CT imaging of 3-D distribution of radiotracer" has been added to improve contrast resolution and lesion placement.

Despite the known greater sensitivity of SPECT compared to planar bone nuclear medicine studies, SPECT is usually done only in limited patients due to time constraints. This is because a standard tomographic bone acquisition requires about 20 minutes, therefore it usually can only be performed over one body region such as the abdomen or chest.

Skeletal PET scanning with F-18 Fluoride has become popular since the introduction of multiple PET scanners for imaging cancer with F-18 FDG. It provides much higher count rates than traditional bone scans done with Tc-99m phosphates, and many authors have shown that it is the most sensitive imaging modality for detecting skeletal lesions. Indeed, several PET centers have proposed replacing the standard Tc-99m bone scan with F-18 PET scans. However the short half-life of F-18 makes this type of study practical only for PET centers within a short distance from a cyclotron. Furthermore, most PET scanners are usually fully occupied doing other types of diagnostic oncology studies, and the cost of the F-18 is currently not reimbursed for simple skeletal surveys.

Recently it has become feasible to dramatically shorten the time necessary for acquisition of a nuclear medicine SPECT study. This has occurred with the introduction of new image reconstruction software which includes resolution recovery correction (so called "collimator de-blurring"). Since this approach results in significant improvement of image resolution, many centers are currently looking at the feasibility of using this new technique to reduce imaging times. For example, its use has been investigated for nuclear cardiac scans with acquisition times shortened by half.

We propose to investigate the performance of the image reconstruction software with resolution recovery correction for bone SPECT studies. We estimate that in only 30 minutes, using this new technique of collimator de-blurring, one could perform a fully 3-dimensional SPECT whole-body bone study, essentially obviating the necessity for doing planar bone studies.

In the scope of the proposed project, our group aims to test the hypothesis that one can perform a Tc-99m whole-body SPECT study in the same time as a regular routine planar bone study, with greater localization accuracy, and greater lesion detection.

To establish a "gold standard" necessary to assess the performance of the SPECT bone scans, we will compare number of malignant lesions detected in patients who are proven to have metastatic skeletal bone lesions on PET F-18 whole-body scans, with whole-body Tc-99m SPECT lesions. We also propose to compare the detection of SPECT scans with standard planar bone scans. This will allow for two major comparisons (a) the accuracy of SPECT bone studies compared to planar bone studies, and (b) the accuracy of SPECT bone scans compared to F-18 PET studies. Most prior studies purporting to show the superiority of F-18 bone scans to Tc-99 bone scans were done only against either planar scans or a combination of planar scans and partial SPECT studies over the spine. We anticipate that F-18 bone scans, due to the higher counting statistics of PET agents, will show more lesions than SPECT, but the exact increase in sensitivity has never been compared to whole-body SPECT scans.

Objectives

1. Evaluate the feasibility of implementing whole-body SPECT in routine practice with standard SPECT gamma cameras
2. Evaluate the value of whole-body SPECT compared to whole-body planar studies for the detection of bone metastases
3. Compare the results of state-of-the art whole-body SPECT skeleton surveys with state-of-the art whole-body Na18F PET whole-body bone surveys.
4. Obtain preliminary data on the respective accuracy of planar bone scintigraphy, whole-body SPECT and Na18F PET/CT to plan future studies on the cost-effectiveness of these methods to improve prostate cancer staging.

Hypotheses

1. A whole-body bone SPECT is more sensitive and specific than a conventional planar bone scan for the detection of bone metastases
2. Whole-body bone SPECT is less sensitive than a whole-body bone PET but the lower sensitivity has minimal impact on the overall detection of bone metastases on a patient basis

Overall study design

This is an open phase II study designed to accumulate preliminary data on the relative diagnostic value of planar bone scintigraphy, whole-body bone SPECT and whole-body bone PET with sodium 18F-Fluoride. We plan to accrue a total of 25 subjects with suspected bone metastases who will undergo planar bone scintigraphy, bone SPECT and a Na18F whole-body bone PET scan.

Data analysis

All patients studies will be analyzed by 3 independent nuclear medicine readers, with number of lesions identified on planar scans being compared to number of lesions on non-Astonish SPECT bone scans and Astonish SPECT bone scans.

Each study will be scored by noting:

* number and localization of lesions detected
* level of certainty (1 = definitely malignant, 5= definitely benign)
* general visual quality of images (graded from 1 = poor to 5 = excellent)

The Na18F PET/CT bone study will serve as the reference gold-standard study against which the other acquisitions will be judged.

Statistical consideration

This is a pilot study which will provide preliminary data for further power calculations to estimate the study size needed to demonstrate a statistically significant improvement of whole-body SPECT compared to planar scintigraphy. With 25 subjects, we will have 82% of chance to demonstrate a statistically significant 30% difference in accuracy between planar scintigraphy and whole-body SPECT compared to the reference standard (PET/CT).

ELIGIBILITY:
Inclusion Criteria:

* Patients with a prior history of prostate cancer and
* clinically suspected bone metastases based on symptoms, radiological examinations or abnormal biochemistry results

Exclusion Criteria:

* Inability to consent to participate in the research study.
* Inability to lie supine for a period of at least 45 minutes.
* Inability to travel to the examination site to undergo the PET/CT examination.
* ECOG/WHO performance status ≥ 2

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Over the last 3-4 months, 60 anonymized patient studies were acquired using concurrent acquisition protocol with 20s, 15s, 10s, and 5s per view and with a total of 64 views (32 views/head). The data from these studies will be used to optimize the reconstruction process and establish the definitive reconstruction parameters to be used in the current study.
  We plan to accrue a total of 25 subjects with suspected bone metastases who will undergo planar bone scintigraphy, bone SPECT and a Na18F whole-body bone PET scan.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2009-01; Primary Completion 2016-08-10 (Actual); Study Completion 2016-08-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anna Celler, PhD, Principal Investigator — University of British Columbia; Philip Cohen, Study Director — University of British Columbia; Francois Benard, Study Director — University of British Columbia
Locations (3):
- Canada (3):
  - Lions Gate Hospital, North Vancouver, British Columbia
  - British Columbia Cancer Agency, Vancouver, British Columbia
  - Vancouver Coastal Health Research Institute, Vancouver, British Columbia